CLINICAL TRIAL: NCT01809821
Title: Sleep to Lower Elevated Blood Pressure: A Randomised Controlled Trial
Brief Title: Sleep to Lower Elevated Blood Pressure
Acronym: SLEPT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College Hospital Galway (Other)
Collaborators: Health Research Board, Ireland (Other)
Responsible Party: Principal Investigator, Dr. Emer McGrath, Dr.Emer McGrath, University College Hospital Galway
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HRBCRFG-150213-EMG
Record Dates: First submitted 2013-03-08; First posted 2013-03-13 (Estimated); Last update posted 2014-09-03 (Estimated); Status verified 2014-09

CONDITIONS: Hypertension; Sleep Disorders; Insomnia; Cardiovascular Diseases
Keywords: Hypertension; Sleep Disorders; Insomnia; Cardiovascular Diseases; Internet treatment
MeSH Terms: conditions — Hypertension; Sleep Wake Disorders; Sleep Initiation and Maintenance Disorders; Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Online Sleep Education (Experimental): The sleep intervention is a multi-component online intervention consisting of sleep information and sleep hygiene education, along with behavioural and cognitive components.
  Interventions: Behavioral: Online Sleep Education
- Usual CV care (No Intervention): Specialist nurses will administer the CV risk factor education intervention to participants in small groups over one hour.

INTERVENTIONS:
Behavioral: Online Sleep Education
  Arms: Online Sleep Education

SUMMARY:
Sleep is an essential component of good physical and mental health. Previous studies have reported that poor quality sleep is associated with an increased risk of hypertension, stroke and cardiovascular disease (CVD). Hypertension is the most common and important risk factor for CVD, and even modest reductions in blood pressure result in significant reductions in stroke and myocardial infarction. In this randomised trial, the investigators aim to evaluate whether a simple, multi-component, online sleep intervention reduces blood pressure in patients with essential hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* ≥18 years on entry to study
* Average automated Systolic Blood Pressure (SBP) monitor readings between 130 - 160 mmHg with average automated Diastolic Blood Pressure(DBP) monitor readings <110 mmHg on three occasions, measured in a valid standardized manner while seated, or average Ambulatory Blood Pressure Monitor (ABPM) SBP reading between 130-160 mmHg with average DBP reading <110 mmHg.
* Self-reported difficulty getting to sleep (defined as usually taking more than 30 mins to get to sleep), and/or staying asleep (usually waking up more than once per night) for at least 3 months duration
* Internet access and self-reported competency in using the internet

Exclusion Criteria:

* Receiving > 2 antihypertensive medications, or recent change in antihypertensive medications (within previous 2 months) or planned change in antihypertensive medication in next 8 weeks
* Previous history of myocardial infarction, ischaemic stroke or transient ischaemic attack
* Previous history of congestive heart failure
* History of dialysis for chronic renal impairment or evidence of chronic kidney disease (eGFR <60 or albuminuria).
* Known history of diabetes mellitus
* Current ongoing sleep hygiene education or sleep related cognitive behavioural therapy
* Ongoing involvement in night shift work
* History of obstructive sleep apnoea (OSA) and previously received or currently receiving treatment for OSA (patients with a history of untreated OSA are eligible for inclusion).
* Known history of sleep disorders (i.e. narcolepsy; hypersomnias; parasomnias such as sleep walking, night terrors, recurring nightmares; periodic limb movements/restless leg syndrome; circadian rhythm sleep disorder)
* Unable to follow educational advice in the opinion of the clinician
* Baby or young children at home that wake during the night
* History of bipolar affective disorder
* History of psychosis
* History of major depression (defined as depression requiring hospitalization in the past or visit to psychiatry outpatient clinic in the past 3 months)
* Unstable depression (unstable will be defined as changes in antidepressant medications within the last 3 months - i.e. start, stop or change in dose.)
* Unstable anxiety disorders/panic attacks (unstable will be defined as changes in medications within the last 3 months - i.e. start, stop or change in dose.)
* Ongoing substance or alcohol abuse
* Planned surgery or hospitalization over the next 8 weeks (i.e. during the trial)
* Incapacitating pain or illness or other medical condition in which, in the opinion of the clinician, the sleep intervention is unlikely to be effective.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2013-05; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Systolic Blood Pressure | 8 weeks
  To determine if the addition of a multi-component, online, sleep intervention to usual care (standard CV risk factor education), results in a greater reduction in mean 24-hr systolic blood pressure in patients with hypertension and poor sleep quality, compared to usual care alone, over an 8-week period.

SECONDARY OUTCOMES:
Diastolic Outcome Measure | 8 weeks
  Is the addition of a multi-component online sleep intervention to usual care (standard CV risk factor education), associated with a greater reduction in mean 24-hr diastolic blood pressure in patients with hypertension and poor sleep quality, compared to usual care alone, over an 8-week period?
Sleep efficiency | 8 weeks
  Change in proportion of participants with sleep efficacy ≥ 85% at 8 weeks
Sleep onset latency | 8 weeks
  Change in proportion of participants with sleep onset latency ≤ 30 minutes at 8 weeks
PSQI | 8 weeks
  Change in proportion of participants with Pittsburgh Sleep Quality Index (PSQI) score <5 over 8 weeks
SCI | 8 weeks
  Change in proportion of participants with sleep condition indicator (SCI) score ≤5.9 at 8 weeks
ISI | 8 weeks
  Change in proportion of participants with Insomnia Severity index (ISI) score ≥15 at 8 weeks

OTHER OUTCOMES:
Body Mass Index | 8 weeks
  Is the addition of a multi-component online sleep intervention to usual care (standard CV risk factor education), associated with greater improvements in body mass index in patients with hypertension and poor sleep quality, compared to usual care alone, over an 8 week period?
Plasma lipoproteins | 8 weeks
  Is the addition of a multi-component online sleep intervention to usual care (standard CV risk factor education), associated with greater improvements in plasma lipids in patients with hypertension and poor sleep quality, compared to usual care alone, over an 8 week period?
Plasma HbA1c | 8 weeks
  Is the addition of a multi-component online sleep intervention to usual care (standard CV risk factor education), associated with greater improvements in plasma HbA1c in patients with hypertension and poor sleep quality, compared to usual care alone, over an 8 week period?
eGFR | 8 weeks
  Is the addition of a multi-component online sleep intervention to usual care (standard CV risk factor education), associated with greater improvements in eGFR in patients with hypertension and poor sleep quality, compared to usual care alone, over an 8 week period?
Insomnia Severity Index | 8 weeks
  Is the addition of a multi-component online sleep intervention to usual care (standard CV risk factor education), associated with greater improvements in Insomnia Severity Index Score in patients with hypertension and poor sleep quality, compared to usual care alone, over an 8 week period?
Sleep Condition Indicator Score | 8 weeks
  Is the addition of a multi-component online sleep intervention to usual care (standard CV risk factor education), associated with greater improvements in Sleep Condition Indicator Score in patients with hypertension and poor sleep quality, compared to usual care alone, over an 8 week period?
Pittsburgh Sleep Quality Index | 8 weeks
  Is the addition of a multi-component online sleep intervention to usual care (standard CV risk factor education), associated with greater improvements in Pittsburgh Sleep Quality Index in patients with hypertension and poor sleep quality, compared to usual care alone, over an 8 week period?
Mean number of cigarettes smoked | 8 weeks
  Is the addition of a multi-component online sleep intervention to usual care (standard CV risk factor education), associated with greater improvements in mean number of cigarettes smoked in patients with hypertension and poor sleep quality, compared to usual care alone, over an 8 week period?
Sleep onset latency | 8 weeks
  Is the addition of a multi-component online sleep intervention to usual care (standard CV risk factor education), associated with greater improvements in sleep onset latency in patients with hypertension and poor sleep quality, compared to usual care alone, over an 8 week period?
Wake time to sleep onset | 8 weeks
  Is the addition of a multi-component online sleep intervention to usual care (standard CV risk factor education), associated with greater improvements in wake time to sleep onset in patients with hypertension and poor sleep quality, compared to usual care alone, over an 8 week period?
Sleep efficiency | 8 weeks
  Is the addition of a multi-component online sleep intervention to usual care (standard CV risk factor education), associated with greater improvements in sleep efficiency in patients with hypertension and poor sleep quality, compared to usual care alone, over an 8 week period?
Beck Depression Inventory score | 8 weeks
  Is the addition of a multi-component online sleep intervention to usual care (standard CV risk factor education), associated with greater improvements in Beck Depression Inventory score in patients with hypertension and poor sleep quality, compared to usual care alone, over an 8 week period?
Beck Anxiety Inventory score | 8 weeks
  Is the addition of a multi-component online sleep intervention to usual care (standard CV risk factor education), associated with greater improvements in Beck Anxiety Inventory score in patients with hypertension and poor sleep quality, compared to usual care alone, over an 8 week period?
Smoking status | 8 weeks
  Is the addition of a multi-component online sleep intervention to usual care (standard CV risk factor education), associated with a change in smoking status compared to usual care alone, over an 8 week period?
Diastolic blood pressure | 8 weeks
  Is the addition of a multi-component online sleep intervention to usual care (standard CV risk factor education), associated with a change in daytime (peak and mean) diastolic blood pressure , compared to usual care alone, over an 8 week period?
Systolic blood pressure | 8 weeks
  Is the addition of a multi-component online sleep intervention to usual care (standard CV risk factor education), associated with a change in daytime (peak and mean) systolic blood pressure , compared to usual care alone, over an 8 week period?
Total Sleep Time | 8 weeks
  Is the addition of a multi-component online sleep intervention to usual care (standard CV risk factor education), associated with a change in Total Sleep Time , compared to usual care alone, over an 8 week period?
Diastolic blood pressure | 8 weeks
  Is the addition of a multi-component online sleep intervention to usual care (standard CV risk factor education), associated with a change in nighttime (peak and mean) diastolic blood pressure , compared to usual care alone, over an 8 week period?
Systolic blood pressure | 8 weeks
  Is the addition of a multi-component online sleep intervention to usual care (standard CV risk factor education), associated with a change in nighttime (peak and mean) systolic blood pressure , compared to usual care alone, over an 8 week period?
Systolic blood pressure | 8 weeks
  Is the level of adherence to a multi-component online sleep intervention associated with a change in mean 24-hour SBP over 8 weeks
Systolic blood pressure | 8 weeks
  To determine if concomitant use of antihypertensive medication influences the change in mean 24-hour SBP over 8 weeks .

CONTACTS AND LOCATIONS:
Overall Officials: Martin J O'Donnell, MB PhD, Principal Investigator — National University of Ireland, Galway
Locations (1):
- HRB Clinical Research Facility Galway, Galway, Ireland

REFERENCES:
- [Derived] McGrath ER, Espie CA, Murphy AW, Newell J, Power A, Madden S, Byrne M, O'Donnell MJ. Sleep to lower elevated blood pressure: study protocol for a randomized controlled trial. Trials. 2014 Oct 9;15:393. doi: 10.1186/1745-6215-15-393. PMID 25300874